CLINICAL TRIAL: NCT00827970
Title: Populationbased Screening for Urogenital Chlamydia Trachomatis Infections by Use of Home-Obtained and Mailed Samples: A Randomized Study
Brief Title: Randomized Population-Based Study on Chlamydia Trachomatis Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus County, Denmark (Other); Novo foundation (Unknown); The Danish Medical Research Council (Other)
Responsible Party: Berit Andersen, MD, Ph.D., Aarhus University Hospital Skejby, Department of Infectious Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Cesoirs01
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Chlamydia Trachomatis; Infertility; Ectopic Pregnancy
Keywords: mass screening
MeSH Terms: conditions — Infertility; Pregnancy, Ectopic | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Screening (Experimental): Individuals receiving an invitation to be tested for urogenital Chlamydia trachomatis by use of a home-obtained and mailed sample.
  Interventions: Behavioral: Screening for urogenital Chlamydia trachomatis
- 2 Control (No Intervention): Control group receiving usual care

INTERVENTIONS:
Behavioral: Screening for urogenital Chlamydia trachomatis — Receeiving an invitation to be tested for urogenital Chlamydia trachomatis by use of a home-obtained and mailed sample.
  Arms: 1 Screening

SUMMARY:
30,000 individuals living in Aarhus County, Denmark by Oct 1997 were randomized into two groups. The intervention group received an invitation to be tested for urogenital Chlamydia trachomatis by use of home-obtained and mailed sample (9,000 individuals). The control group received no intervention (21,000 individuals). Outcome measures: Number of tested individuals, number of detected infections, number of women developing PID, ectopic pregnancy or infertility, number of women giving birth to a child, number of women receiving IVF treatment and number of men developing epididymitis.

The hypothesis was that more individuals would be tested and treated for infections and that number of long term fertility complications would decline in the intervention group compared to control group.

ELIGIBILITY:
Inclusion Criteria:

* born in 1974, 1974 or 1976 AND living in Aarhus County October 1007

Exclusion Criteria:

-

Ages: 21 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30000 (Actual)
Dates: Start 1997-10; Primary Completion 1998-02 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Long term infertility complications | 2008

CONTACTS AND LOCATIONS:
Overall Officials: Berit Andersen, MD, Ph.D., Principal Investigator — Aarhus University Hospital Skejby, Department of Infectious Diseases
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital Skejby, Aarhus N, Denmark

REFERENCES:
- [Result] Andersen B, Olesen F, Moller JK, Ostergaard L. Population-based strategies for outreach screening of urogenital Chlamydia trachomatis infections: a randomized, controlled trial. J Infect Dis. 2002 Jan 15;185(2):252-8. doi: 10.1086/338268. Epub 2002 Jan 3. PMID 11807700
- [Derived] Andersen B, van Valkengoed I, Sokolowski I, Moller JK, Ostergaard L, Olesen F. Impact of intensified testing for urogenital Chlamydia trachomatis infections: a randomised study with 9-year follow-up. Sex Transm Infect. 2011 Mar;87(2):156-61. doi: 10.1136/sti.2010.042192. Epub 2010 Nov 20. PMID 21097811